CLINICAL TRIAL: NCT05479760
Title: Key Population-Led Same Day Test and Treat for Hepatitis C in Community-Based Organizations in Bangkok, Thailand: A Demonstration Project
Brief Title: KP-Led Same Day HCV Test and Treat Study
Acronym: 479/65
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IHRI018
Record Dates: First submitted 2022-07-06; First posted 2022-07-29 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-11

CONDITIONS: HCV, HIV
Keywords: HCV, HIV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation for anti-HCV reactive client (Experimental): All clients who test anti-HCV positive at the study CBOs will be assessed for the inclusion criteria. Eligible clients will be informed and offered to participate in the study.
  Interventions: Other: KP-Led HCV test and treat service

INTERVENTIONS:
Other: KP-Led HCV test and treat service — After completing informed consent procedures, screening procedures will take place to assess eligibility. Clients who are anti-HCV and HCV-RNA positive, but meet one/more ineligible characteristics for simplified treatment will be referred to a hepatologist for treatment initiation.
  Participants who are HCV-RNA positive and otherwise eligible will be offered to initiate DAAs at the CBO, followed by telehealth visits at week 4 and 8 and CBO visits at week 12, and week 24. If a visit is requested by the client, it can be conducted through telehealth or in-person at the clinic depending on client preferences. Substance use will be assessed using ASSIST, Retention in care, occurrence of adverse events during treatment, completion of treatment, and SVR achievement will be assessed. Clients who achieve SVR will be retested with HCV-RNA every 3 months to assess HCV re-infection. Clients who do not achieve SVR will be referred for further analysis and treatment.

SUMMARY:
This is a Hybrid design to primarily assess effectiveness, and to secondarily observe and collect data on the implementation of the service. This will allow the assessment of health-related outcomes and implementation outcomes to facilitate dissemination and replication if proven to be successful in other CBOs in Thailand, regionally, and globally.

DETAILED DESCRIPTION:
Implementation Effectiveness To assess effectiveness, an interrupted time series (ITS) design. The counterfactual scenario (under which KP-led HCV test and treat had not been implemented) will be determined using routine service data collected from 15 months prior to the study implementation, and will provide a comparison for the evaluation of the impact of KP-led HCV test and treat by examining any change occurring in the primary outcomes in the post-implementation period during the 15 months of the study.

Implementation Strategies To assess implementation, Proctor's model was used to guide the selection of relevant implementation outcomes, which during this stage of implementation are acceptability, feasibility, and fidelity. Socio-ecological level, framework, and relevant constructs for each outcome are outlined below and in table 1.

1. Acceptability of KP-led HCV test and treat Acceptability refers to the perception that the service is agreeable and satisfactory. It will be measured using surveys at four socio-ecological levels, informed by different frameworks according to relevance

   * Clients, pre-implementation: The Health Belief Model (HBM) will be used to design a survey to assess determinants that drive the acceptability of HCV test and treat services at the CBO. The HBM is one of the first theories of health behavior, and addresses the individual's perception of the threat posed by a health problem and factors influencing the decision to act. This assessment will be conducted pre-implementation, and findings will inform the design of implementation strategies targeting clients
   * Clients, during implementation: To assess the acceptability and satisfaction of the same day HCV test and treat service, clients who initiated DAA treatment at the CBO will be asked to complete a standard survey on acceptability and satisfaction
   * Providers: The Theory of Planned Behavior (TPB) will be used to design a survey to assess factors that influence the acceptability of HCV test and treat among KP-lay providers. The TPB examines the relations between an individual's belief, attitudes, intentions, behavior, and perceived control over that behavior. This assessment will be conducted pre-implementation, and findings will inform the design of implementation strategies targeting providers.
   * CBO leadership: The Theory of Planned Behavior (TPB) will also be used to design a survey to assess factors that influence the acceptability of HCV test and treat among CBO leaderships. This assessment will be conducted pre-implementation, and findings will inform the design of implementation strategies targeting CBO leadership.
   * Policy makers: The Consolidated Framework for Implementation Research (CFIR) will be used to produce interview guides to assess the acceptability of the service among key government stakeholders and policy makers.
2. Feasibility of providing KP-led HCV test and treat by KP-lay providers in CBOs

   Feasibility refers to the extent to which the service can be successfully delivered within the CBO setting. It will be measured at two socio-ecological levels:
   * Providers: Training records, and surveys and in-depth interviews informed by CFIR.
   * CBO leadership: CFIR will be used to design surveys to assess relevant domains and constructs, and in-depth interviews will be conducted to further explore survey findings.
3. Fidelity of KP-led HCV test and treat implementation Fidelity refers to the extent to which the service was delivered as intended. It will be measured at the provider level using observation, checklists, and assessment of client records, guided by CFIR.

ELIGIBILITY:
Eligibility criteria for assessment of effectiveness outcomes:

Inclusion Criteria:

* Thai citizen
* 18 years or older
* Signed informed consent
* Tested anti-HCV positive

Exclusion Criteria:

* Decline to participate in the research

Eligibility criteria assessment of implementation outcomes:

Inclusion criteria:

* Client level: Tested anti-HCV positive at one of the implementing CBOs
* Provider level: KP lay providers providing KP-led Same Day HCV Test and Treat
* Leadership level: leadership of implementing CBOs
* Government level: involved in policy making related to HCV testing and treatment in key populations

Exclusion criteria:

* Do not provide informed consent to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
The proportion of eligible clients initiating DAAs | 18 months
  The proportion of eligible clients initiating DAAs in CBOs under KP-led HCV test and treat in CBOs as compared to pre-implementation.
The proportion of complete tretmented client | 18 months
  The proportion of clients who complete 12 weeks of treatment under KP-led HCV test and treat in CBOs as compared to pre-implementation.
The proportion of SVR achieved client | 18 months
  The proportion of clients who achieve SVR at 12 weeks after treatment completion under KP-led HCV test and treat in CBOs as compared to pre-implementation.

SECONDARY OUTCOMES:
The HCV re-infection rates | 18 months
  Proportion of clients with HCV-reinfection among those who had previously achieved SVR
The duration to DAA initiation among clients with chronic HCV infection | 18 months
  Time from anti-HCV positivity to DAA initiation among clients with chronic HCV infection pre- compared to post-implementation
The acceptability of KP-led HCV test and treat | 18 months
  The acceptability of KP-led HCV test and treat will be measured via survey and/or in-depth interviews with clients, providers, CBO leadership, and policymakers
Provider perception of KP-led HCV test and treat feasibility. | 18 months
  The feasibility of providing KP-led HCV test and treat will be measured via survey and/or in-depth interviews with KP-lay providers.
The fidelity of provider during the implementation | 18 months
  The KP-led HCV test and treat fidelity of KP-lay providers will be assessed through service delivery checklists and case report forms.

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Rainbow Sky Association of Thailand (RSAT), Bangkok, Bangkapi
  - Institute of HIV Research and Innovation, Pathum Wan, Bangkok
  - The Service Workers In Group Foundation (SWING), Bangkok, Building 3, Patpong, Surawong Road
  - MPLUS Foundation (MPLUS), Chiang Mai